CLINICAL TRIAL: NCT02020148
Title: Can Prenatal Plasma Oxytocin Concentration Predict Likelihood of Postpartum Depression? An Opportunity for Early Intervention and Prevention in a Vulnerable Population
Brief Title: Can Oxytocin Level Predict Postpartum Depression?
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Northwestern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 00082402
Record Dates: First submitted 2013-12-12; First posted 2013-12-24 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Postpartum Depression
Keywords: pregnancy; oxytocin; postpartum depression; depression; pregnant women; mood; anxiety; hormones; women's health; mental health; baby blues; mood disorders
MeSH Terms: conditions — Depression, Postpartum; Depression; Anxiety Disorders; Psychological Well-Being; Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A 3 milliliter (about half a teaspoon) blood sample will be obtained to measure oxytocin level.
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this research study is to understand the relationship between the hormone oxytocin and postpartum mood.

DETAILED DESCRIPTION:
Postpartum depression (PPD) affects some one in five new mothers, and adversely influences maternal adaptation to motherhood. While it is known that women with a prior history of depression, or depression during pregnancy, are at elevated risk for postpartum depression, many women with no prior history of depression or other risk factors go on to develop depression in the postpartum period. Considering the grave consequences of postpartum depression on maternal infant bonding and childhood psychological development, it is critical to develop reliable methods to identify which women, who are not depressed during pregnancy, will become depressed after delivery.

The biological pathways leading to depression at any time in life, including around pregnancy, are still poorly characterized. Oxytocin (OT), a hormone involved in delivery and lactation, has received recent attention regarding its additional role in maternal emotions and care taking behaviors after birth. The primary goal is explore the relationship between plasma oxytocin and postpartum mood.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. English-speaking
3. Pregnant (third trimester at time of visit)

Exclusion Criteria:

1. Current active depression or other mental illness at time of study entry in the third trimester (past depression or anxiety is acceptable)
2. Current antidepressant treatment
3. Severe medical complications in current pregnancy (gestational diabetes, hypertension, thyroid disease)
4. Signs of multiple gestation or of fetal malformation in current pregnancy
5. Cigarette smoking beyond 10th week of gestation of current pregnancy
6. Pre-pregnancy BMI > 32

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Pregnant Women
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Inventory of Depressive Symptomatology, Self-Report (IDS-SR-30) | 4-6 weeks post delivery
  The IDS-SR-30 is a validated, widely used tool to evaluate depressive symptoms and clinical depression. Participants will complete this questionnaire in person or through telephone interview.

CONTACTS AND LOCATIONS:
Overall Officials: Suena H Massey, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Result] Bell AF, Carter CS, Steer CD, Golding J, Davis JM, Steffen AD, Rubin LH, Lillard TS, Gregory SP, Harris JC, Connelly JJ. Interaction between oxytocin receptor DNA methylation and genotype is associated with risk of postpartum depression in women without depression in pregnancy. Front Genet. 2015 Jul 21;6:243. doi: 10.3389/fgene.2015.00243. eCollection 2015. PMID 26257770
- See also: Reference citation — https://www.frontiersin.org/articles/10.3389/fgene.2015.00243/full